CLINICAL TRIAL: NCT00932464
Title: An Open-Label, Randomized, Single-Dose, 2-Period Crossover Study To Determine The Effect Of A High-Fat Meal On The Relative Bioavailability And Pharmacokinetics Of A Single Dose Of The 240 mg Formulation Of Neratinib In Healthy Subjects
Brief Title: Study Evaluating The Effect Of A High-Fat Meal On The Pharmacokinetics Of Neratinib
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study withdrawn as it no longer is deemed necessary per project status.
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3144A2-1112; B1891007
Record Dates: First submitted 2009-07-01; First posted 2009-07-03 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
MeSH Terms: interventions — neratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Neratinib Fasted
  Interventions: Drug: Neratinib
- 2 (Experimental): Neratinib Fed
  Interventions: Drug: Neratinib

INTERVENTIONS:
Drug: Neratinib — 240-mg oral tablet; single dose under fasted conditions
  Other Names: HKI-272
  Arms: 1
Drug: Neratinib — 240-mg oral tablet; single dose with high-fat breakfast
  Other Names: HKI-272
  Arms: 2

SUMMARY:
This study is being conducted to see if neratinib is absorbed, distributed, or eliminated differently when administered in the fasting state versus after a high-fat meal.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women of nonchildbearing potential, age 18 to 50 years.

Exclusion Criteria:

* Any previous or current clinically significant medical condition or disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics as measured by AUC, Cmax, tmax, t1/2 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology